CLINICAL TRIAL: NCT03612791
Title: Randomized Phase II Trial Assessing the Inhibitor of Programmed Cell Death Ligand 1 (PD-L1) Immune Checkpoint Atezolizumab in Locally Advanced Cervical Cancer
Brief Title: Trial Assessing the Inhibitor of Programmed Cell Death Ligand 1 (PD-L1) Immune Checkpoint Atezolizumab
Acronym: ATEZOLACC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003622-33; 2017/2608 (Other: CSET number)
Record Dates: First submitted 2018-07-20; First posted 2018-08-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — atezolizumab; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Treatment Arm (Active Comparator): Radiotherapy (RT):
  * Pelvic +/- para-aortic EBRT (IMRT): 45 Gy in 25 fractions over 5 weeks (Weeks 1-5, with simultaneously integrated boosts to macroscopically involved lymph nodes, if any, in order to deliver a total dose of 60 Gy to macroscopic lymph nodes (including the dose delivered by brachytherapy).
  * Uterovaginal brachytherapy (Week 7; maximum interval between EBRT and brachytherapy: 14 days). If appropriate and feasible, dose escalation will be assumed, particularly for advanced disease, with the objective to deliver a minimal total dose of 85 Gy (equivalent dose in 2-Gy fractions with α/β=10 Gy) to 80% of the High Risk-Clinical Target Volume (HR-CTV), including 45 Gy through EBRT. The total dose might be lower in case of close proximity to organs at risk (OARs).
  * Total duration of RT (including brachytherapy) should be ≤ 55 days.
  Chemotherapy:
  - Cisplatin infused 40 mg/m2 (maximum 70 mg) weekly IV during EBRT (Weeks 1-5).
  Interventions: Radiation: Radiotherapy; Drug: Cisplatin
- Experimental Treatment Arm (Experimental): * Same treatment as described above (CRT, followed by uterovaginal brachytherapy), plus
  * atezolizumab administered IV 1200 mg Q3W, starting on the same week as EBRT (Week 1) and continued as an adjuvant for a total maximum of 20 cycles (approximately 14 months total of treatment).
  Interventions: Drug: Atezolizumab; Radiation: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Atezolizumab — atezolizumab administered IV 1200 mg Q3W, starting one week before EBRT (Week -1) and continued as an adjuvant for a total maximum of 20 cycles.
  Arms: Experimental Treatment Arm
Radiation: Radiotherapy — * Pelvic +/- para-aortic EBRT (IMRT): 45 Gy in 25 fractions over 5 weeks (Weeks 1-5, with simultaneously integrated boosts to macroscopically involved lymph nodes, if any, in order to deliver a total dose of 60 Gy to macroscopic lymph nodes (including the dose delivered by brachytherapy).
  * Uterovaginal brachytherapy (Week 7; maximum interval between EBRT and brachytherapy: 14 days). If appropriate and feasible, dose escalation will be assumed, particularly for advanced disease, with the objective to deliver a total dose of 85 Gy (equivalent dose in 2-Gy fractions with α/β=10 Gy) to 80% of the High Risk-Clinical Target Volume (HR-CTV), including 45 Gy through EBRT. The total dose might be lower in case of close proximity to organs at risk (OARs).
  * Total duration of RT (including brachytherapy) should be ≤ 55 days.
Drug: Cisplatin — * Cisplatin infused 40 mg/m2 (maximum 70 mg) weekly IV during EBRT (Weeks 1-5).
  * Not administered: during the interval between EBRT and brachytherapy, or during brachytherapy, or if radiotherapy is interrupted.

SUMMARY:
The primary objective of this randomized phase II trial is to evaluate the clinical benefits of the addition of atezolizumab to standard chemoradiotherapy (CRT) (first given concurrently with CRT, then continued as adjuvant treatment), compared with CRT alone, on investigator-assessed progression-free survival (PFS), as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (after informing the patient).
2. Age ≥18 years old. Patients above 70 years old will be screened according to the G-8 screening tool. If required (G-8 score ≤14), a consultation with an onco-geriatrician will be held in order to confirm the patient eligibility
3. Histologically confirmed cancer of the uterine cervix: squamous cell carcinoma (SCC), adenocarcinoma, or adenosquamous carcinoma.
4. At least one evaluable lesion according to RECIST v1.1 criteria for the assessment of the principal judgment criteria. At baseline, lesion(s) must be ≥10 mm in the longest diameter (except lymp nodes which must have a short axis ≥15 mm).
5. International Federation of Gynecology and Obstetrics (FIGO 2009) classification (confirmed by both clinical staging and/or imaging):

   (i) stage IB1-IIA tumour with positive pelvic nodal status, as assessed by magnetic resonance imaging (MRI) and/or fluorine-18 fluorodeoxyglucose positron emission tomography (18-FDG PET)/computerised tomography (CT); (ii) stage IIB-IVA tumour, regardless of pelvic lymph node involvement; (iii) stage IVB tumours only if the metastases are limited to the paraaortic lymph nodes.

   No evidence of metastatic disease outside the para-aortic area by primary staging (including clinical examination, pelvic MRI, 18-FDG PET, +/- laparoscopic para-aortic lymph node staging).
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
7. Adequate haematologic and end-organ function, defined by the following laboratory results obtained within 15 calendar days prior to the first study treatment:

   1. Absolute neutrophil count (ANC) ≥1,500/mm3 (≥1.5 x 10^9/L) without granulocyte colony-stimulating factor (G-CSF) support.
   2. Total white blood cells (WBC) >2,000/mm3 (>2.0 x 10^9/L) (including Polymorphonuclear neutrophils > 1,500/mm3 or 1.5 x 10^9/L)
   3. Lymphocyte count ≥500/mm3 (≥ 0.5 x 10^9/L)
   4. Platelet count ≥ 100,000/mm3 (≥ 100 x 10^9/L) without transfusion.
   5. Haemoglobin ≥ 9.0 g/dL (90 g/L; patients may be transfused to meet this criterion).
   6. International Normalized Ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × upper limit of normal (ULN) for patients not receiving therapeutic anticoagulation.

      Patients receiving therapeutic anticoagulation should be on a stable dose.
   7. Creatinine <1.5 ULN or calculated creatinine clearance (CrCL) ≥ 45 mL/min (calculated using the Cockcroft-Gault formula).
   8. Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase <2.5 x ULN.
   9. Serum bilirubin <1.5 x ULN.
8. Proteinuria < 200 mg/dL (2 g/L). Patients with ureteral stent or with bladder invasion are eligible if the proteinuria is above the former threshold
9. Ability to comply with the study protocol.
10. Geographical, social and psychological ability to undergo the followup required by the study.
11. Women who are not postmenopausal (≥ 12 months of non-therapy induced amenorrhoea) and not surgically sterile:

    1. Must agree to either use an acceptable contraceptive method* or to remain abstinent** (refrain from heterosexual intercourse) during the treatment period and for at least 5 months after the last dose of atezolizumab in arm B and at least 6 months after the last cisplatin/carboplatin dose in arm A.

       * Acceptable contraceptive methods include single or combined contraceptive methods that result in a failure rate of < 1% per year, such as: tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.

       ** Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Must have a negative serum pregnancy test result within 7 days prior to initiation of study drug.
12. Patients must be affiliated to a social security system or beneficiary of the same, as per local regulatory requirements

Exclusion Criteria:

1. Histological types of cervical cancer other than those listed in the inclusion criteria (based on FIGO 2009 classification), including:

   1. Stage IB1 and IIA cervical cancer with no regional lymph node metastases (N0).
   2. Stage IVB cervical cancer with presence of distant metastases other than para-aortic lymph node metastases.
2. Prior surgery for cervical cancer unless cone resection and paraaortic lymphadenectomy.
3. Prior pelvic radiotherapy, other radiotherapy, chemotherapy or immunotherapy.
4. Any malignancy other than the disease under study in the past 5 years excepting skin cancers such as BCC or SCC.
5. Pregnant or lactating women, or intending to become pregnant during the study.
6. For patient ≥ 70 years old with a G-8 score ≤ 14, unconfirmation of patient eligibility done by the onco-geriatrician at screening
7. History of clinically relevant cardiovascular disease, congestive heart failure (New York Heart Association [NYHA] Class II or greater), or a known left ventricular ejection fraction (LVEF) <50%, symptomatic coronary artery disease, poorly controlled cardiac arrhythmia, or myocardial infarction.
8. Active inflammatory bowel disease, lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome.
9. Serious infection requiring oral or IV antibiotics within 4 weeks prior to randomisation, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
10. Treatment with another investigational therapy within 30 days prior to initiation of the study drug.
11. Major surgical procedure within 4 weeks prior to randomisation or anticipation of the need for a major surgical procedure during the study other than for diagnosis. The following are not considered a major surgical procedure and are therefore permitted:

    (i) placement of central venous access catheter(s) (e.g., port or similar); (ii) surgical lymph node staging with no perioperative complications; (iii) placement of ureteral catheters.
12. History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.
13. Known hypersensitivity to Chinese hamster ovary (CHO) cell products or any component of the atezolizumab formulation.
14. Any contraindication to the use of Cisplatin and/or carboplatin
15. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, meningoencephalitis, or glomerulonephritis (see Appendix 6 for a more comprehensive list of autoimmune diseases) with the following exceptions: patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, patients with controlled Type 1 diabetes mellitus on a stable insulin regimen, and patients with mild autoimmune skin disorders (such as eczema or atopic dermatitis involving <10% of the skin) may be eligible for this study.
16. History of idiopathic pulmonary fibrosis (IPF, including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or active pneumonitis.
17. Pre-existing hearing impairment.
18. Peripheral neuropathy ≥grade 2
19. Positive test for human immunodeficiency virus (HIV).
20. Active hepatitis B (positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C (positive hepatitis C virus antibody [HCVAb] test at screening). Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antibody [HBcAb] test) are eligible.
21. Known active tuberculosis.
22. Receipt of a live, attenuated vaccine within 4 weeks prior to randomisation or anticipation that such a live, attenuated vaccine will be required during the study. Note: Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist®) within 28 days prior to randomisation, during treatment or within 5 months following the last dose of atezolizumab.
23. Prior treatment with CD137 agonists, anti-PD-1, or anti-PD-L1 therapeutic antibody or immune checkpoint targeting agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | from randomization to the first documented occurrence of disease progression, as determined by the investigator using RECIST v1.1, or death from any cause, whichever occurs first, up to 24 months
  The primary endpoint is progression free survival (PFS), defined as the time from randomization to the first documented occurrence of disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided